CLINICAL TRIAL: NCT00171379
Title: Open-label Study to Evaluate the Tolerability, Safety and Efficacy of the Equimolar Conversion From Mycophenolate Mofetil (MMF) to Enteric-Coated Mycophenolate Sodium (EC-MPS) in Patients With Renal Transplant
Brief Title: Clinical Study to Evaluate the Tolerability, Safety and Efficacy of Enteric-coated Mycophenolate Sodium After Equimolar Conversion From Mycophenolate Mofetil (MMF) in Patients With Renal Transplant
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Novartis External Affairs, Novartis Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CERL080AIT01
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2011-02-02 (Estimated); Status verified 2011-02

CONDITIONS: Prevention of Acute Rejection After Kidney Transplantation
Keywords: Kidney transplantation; acute rejection; gastrointestinal adverse events; quality of life; mycophenolate sodium.

INTERVENTIONS:
Drug: Enteric-Coated Mycophenolate Sodium

SUMMARY:
The aim of the study is to evaluate the safety and efficacy of equimolar conversion from MMF to enteric-coated mycophenolate sodium, in renal transplant patients receiving cyclosporine.

ELIGIBILITY:
Inclusion Criteria:

* First or second (single or double) deceased or living donor kidney transplant received at least six months previously;

  * Immunosuppressive therapy with cyclosporin and mycophenolate mofetil (MMF);
  * Receiving an MMF dose of <2/g/day because of any adverse event and/or altered laboratory test result attributed to MMF

Exclusion Criteria:

* • Subjects expected to discontinue cyclosporin therapy;

  * Patients with thrombocytopenia (<75,000/mm3), an absolute neutrophil count of <1,500/mm3 and/or leukopenia (<2,500/mm3), or anemia (hemoglobin <6 g/dl) at baseline;
  * Patients experiencing an acute rejection in the previous two months, with inadequate (creatininemia >2.5 mg/dL) or worsening renal function in the previous two months.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2004-03; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Renal function, measured as calculated creatinine clearance according to the Cockcroft and Gault formula

SECONDARY OUTCOMES:
Incidence of biopsy proven acute rejection
Overall Gastrointestinal disturbances as measured by visual analog scales (upper and lower gastrointestinal symptoms)
Quality of life related to GI symptoms (GIQLI scale)
Full blood count
Gastrointestinal Adverse Events (check-list)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis